CLINICAL TRIAL: NCT05207111
Title: Single-Dose Fasting Bioavailability Study of Mylan's Revefenacin Inhalation Solution, 175 mcg/3 mL in Healthy Chinese Adult Male and Female Volunteers
Brief Title: Fasting Bioavailability Study of Mylan's Revefenacin Inhalation Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharma UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVE-1-19142
Record Dates: First submitted 2021-09-15; First posted 2022-01-26 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers Bioavailability Study
MeSH Terms: interventions — revefenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Revefenacin Inhalation Solution, 175 mcg/3 mL (Experimental)
  Interventions: Drug: Revefenacin Inhalation Solution

INTERVENTIONS:
Drug: Revefenacin Inhalation Solution — Revefenacin Inhalation Solution, 175 mcg/3 mL following a single nebulized inhaled 175 mcg (1 x 175 mcg/3 mL) dose administered under fasting conditions.
  Other Names: Yupelri

SUMMARY:
Single-Dose Fasting Bioavailability Study of Revefenacin Inhalation Solution, 175 mcg/3 mL in 24 Healthy Chinese Adult Male and Female Volunteers. This study will evaluate the safety and tolerability of Revefenacin Inhalation Solution in the Chinese population. For the determination of the pharmacokinetic disposition of the formulations, The bioavailability of Revefenacin Inhalation Solution, 175 mcg/3 mL will be assessed through various pharmacokinetic parameters derived from the plasma concentration-time curves of revefenacin and its active metabolite, THRX-195518.

DETAILED DESCRIPTION:
A single-dose, open-labeled, one-period, one-treatment study to investigate the bioavailability of Revefenacin Inhalation Solution, 175 mcg/3 mL following administration of a single, nebulized, inhaled 175 mcg (1 x 175 mcg/3mL) dose in a total of 24 healthy, Chinese, adult male and female volunteers under fasting conditions. In addition, this study will evaluate the safety and tolerability of Revefenacin Inhalation Solution in the Chinese population. Ten milliliter (1 × 10 mL) blood samples will be collected at pre-dose and the following times after the initiation of dosing: 5, 10, 15, 30, and 45 minutes along with 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours.

The bioavailability of Revefenacin Inhalation Solution, 175 mcg/3 mL will be assessed through various pharmacokinetic parameters (such as AUC0-t, AUC0-∞, Cmax, and Tmax) derived from the plasma concentration-time curves of revefenacin and its active metabolite, THRX-195518.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Healthy male and female volunteers aged 18 to 55
* Males and/or non-pregnant, non-lactating females.

  1. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

     1. Postmenopausal with spontaneous amenorrhea for at least one (1) year, or spontaneous amenorrhea for less than one (1) year with serum FSH levels >40mIU/ml as confirmed by lab test at screening, or
     2. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
     3. Total hysterectomy and an absence of bleeding for at least 3 months.
  2. Women of childbearing potential will need to have a negative serum β-HCG pregnancy test performed within 14 days prior to the start of the study.
* Weight at least 50 kg (110 lbs) for men and 45 kg (99 lbs) for women and have a Body Mass Index (BMI) value less than or equal to 26.0 kg/m2 but greater than or equal to 19.0 kg/m2.
* Smoking Status: Non-nicotine users only.
* Adequate venous access in both arms for the collection of a number of blood samples during the study.
* Utilization of illiterate subjects is permitted when performed according to GCP, as well as regulations/guidance for the region of submission and country of conductance.
* Willing to follow the protocol requirements and comply with protocol restrictions.
* Negative chest X-ray for tuberculosis may be performed (within 6 months of study and documentation available) at the discretion of the Principal Investigator or Medical Sub Investigator.
* Normal spirometry assessment (FEV1 ≥ 80% predicted and FEV1/FVC ≥ 0.7).
* Negative urine drug screen including at a minimum amphetamines, benzodiazepines, cannabinoid, cocaine, and opiates.
* Negative Rapid Plasma Reagin (RPR, syphilis test) or Venereal Disease Research laboratory (VDRL) test. Tests for other sexually transmitted diseases (STD).
* Subjects should be judged by the Principal Investigator or Medical Sub- Investigator as normal and healthy during a pre-study medical evaluation performed within 14 days of the initial dose of study medication

Exclusion Criteria:

1. Institutionalized subjects.
2. Social Habits

   1. Ingestion of any alcoholic beverage within the 48 hours prior to the initial administration of study medication.
   2. Ingestion of any caffeine- or xanthine-containing food or beverage within the 24 hours prior to the initial administration of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial administration of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. History of drug and/or alcohol abuse within one year of start of study.
   6. Use of any nicotine containing product(s) within 1 year of the initial dose of study medication.
3. Medications

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial administration of study medication.
   2. Use of any hormone replacement therapy within 3 months prior to initial administration of study medication.
   3. A depot injection or implant of any drug within 3 months prior to initial administration of study medication.
   4. Use of any medication, herbal supplement, or vitamin known to induce or inhibit hepatic enzyme activity or transporters within 28 days prior to the initial administration of study medication. (see https://go.usa.gov/xXY9C).
4. Use of any food (e.g. broccoli, Brussels sprouts, char-grilled meat, star fruit, pomegranate, seville oranges grapefruit, grapefruit-like, or grapefruit containing products) known to induce or inhibit hepatic enzyme activity must be limited to no more than 2 standard servings (e.g. one standard serving of char-grilled meat is approximately 12 ounces; one standard serving of vegetables/fruits is approximately 1 cup) per week within 4 weeks prior to the initial dose of study medication. These foods must be discontinued at least 7 days prior to the initial dose of study medication, during the study and until the end of the study.
5. Diseases

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, genitourinary, musculoskeletal disease or malignancies unless deemed not clinically significant by the Principal Investigator or Medical Sub-Investigator
   2. History of tuberculosis.
   3. History of pulmonary problems, such as but not limited to asthma, bronchospasms, and COPD.
   4. Acute illness at the time of either the pre-study medical evaluation or dosing.
   5. History of glaucoma.
   6. History of urinary retention.
   7. History of bladder neck obstruction
   8. History of symptomatic benign prostatic hyperplasia
   9. History of chronic constipation
   10. History of long QT syndrome or Subject has an abnormal ECG at Screening or Day -1, including QT interval corrected for heart rate (HR) using Fridericia's formula (QTcF) >470 milliseconds (msec) (applicable for any screening or baseline ECG), or subject has any cardiac rhythm other than sinus rhythm that is interpreted by the investigator to be clinically significant. All ECGs must be not clinically significant to qualify for enrollment into the study.
6. Any reason which, in the opinion of the Principal Investigator or Medical Sub- Investigator would prevent the subject from safely participating in the study.
7. Intolerance to venipuncture.
8. Donation or loss of blood or plasma: 50 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication.
9. Subjects who have received an investigational drug within 90 days prior to the initial dose of study medication.
10. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Medical Sub-Investigator, could contraindicate the subject's participation in this study.
11. Allergy or hypersensitivity to Revefenacin, other related products, or any inactive ingredients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 0 to 96 hours post-dose
  The maximum concentration (CPEAK)
Bioavailability | 0 to 96 hours post-dose
  The Area under the plasma concentration-time curve (AUCL)
Bioavailability | 0 to 96 hours post-dose
  The time at which it occurred relative to the administered dose (TPEAK)
Bioavailability | 0 to 96 hours post-dose
  Area under the plasma concentration-time curve from zero to infinity (AUCINF)
Bioavailability | 0 to 96 hours post-dose
  The elimination rate constant (KEL)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shaw, PhD, Study Director — Head of Global PKDM Science Oversight
Locations (1):
- Xuzhou Central Hospital, Xuzhou, China

IPD SHARING:
Plan to Share IPD: Undecided